CLINICAL TRIAL: NCT01967641
Title: Prescription Opioid Abuse Among Pain Patients: Predictors of Relapse
Acronym: PAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Frances R Levin, Director of Substance Use Disorder, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #6269R; DA020448-05 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Opioid Dependence
Keywords: opioid dependence; opioid abuse; suboxone; prescription pain medications
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Masking Description: Following induction, patients were stabilized beginning on Day 2 on one of three blinded doses of buprenorphine/naloxone (2/0.5, 8/2, or 16/4 mg per day) for a week then underwent laboratory testing for a second week. Each blinded buprenorphine dose was administered in equal divided doses according to a QID dosing schedule, and each dose was maintained for a two-week period, with the second week including laboratory testing.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- buprenorphine/naloxone combination (Experimental): Buprenorphine/naloxone (Bup/Nx; Suboxone sublingual tablets, Reckitt Benckiser) will be administered sublingually at daily doses of 2/0.5, 8/2 mg, and 16/4 mg, which are within the recommended dose range for treating both pain and opioid abuse. The total daily dose will be divided and administered on a QID dosing regimen (0.5/0.125, 2/0.5, and 4/1 mg QID at 0830, 1230, 1730, 2130). Each participant will be tested with all three doses in random order for two weeks at each dose (one week of stabilization followed by one week of testing). Following completion of the 7-week inpatient phase, participants will be followed at the Substance Use Research Center (SURC) and maintained on 16/4 mg Bup/Nx.
  Interventions: Drug: buprenorphine/naloxone combination

INTERVENTIONS:
Drug: buprenorphine/naloxone combination — Buprenorphine/naloxone (Bup/Nx; Suboxone sublingual tablets, Reckitt Benckiser) will be administered sublingually at daily doses of 2/0.5, 8/2 mg, and 16/4 mg, which are within the recommended dose range for treating both pain and opioid abuse. The total daily dose will be divided and administered on a QID dosing regimen (0.5/0.125, 2/0.5, and 4/1 mg QID at 0830, 1230, 1730, 2130). Each participant will be tested with all three doses in random order for two weeks at each dose (one week of stabilization followed by one week of testing). Following completion of the 7-week inpatient phase, participants will be maintained on 16/4 mg Bup/Nx.
  Other Names: Suboxone

SUMMARY:
In this study, we will assess opioid self-administration in a laboratory setting in persons with pain who have a history of opioid abuse. Participants diagnosed with mild to moderate pain will be admitted to hospital for 7 weeks and transitioned from their baseline prescription opioid to a standing daily dose of Suboxone (buprenorphine/naloxone combination). During this maintenance period, participants will have the opportunity in a laboratory setting to self-administer oxycodone; subjective responses as well as analgesic, physiological and performance effects will be measured. In the second phase of this study, the same patients who participated in the inpatient phase will be followed on an outpatient basis while maintained on Suboxone for 12 weeks. . The hypotheses of this study are that (1) higher progressive ratio break-point values for oxycodone, higher subjective ratings of euphoria, and less pain relief will predict early relapse to opioid abuse; (2) the abuse liability measures will be more strongly correlated with relapse than the pain measures; (3) subjective ratings of euphoria will increase and of pain will decrease in an oxycodone dose-dependent manner (i.e. euphoria will increase and pain will decrease as dose increases); and (4) experimentally induced pain will decrease in an oxycodone dose-dependent manner.

DETAILED DESCRIPTION:
All participants will be admitted to the GCRU, the SRU, or the CRR and maintained on sublingual Bup/Ntx. During the first week after admission, participants will be withdrawn from their prior opioid analgesic regimen and will be stabilized on one of three doses of buprenorphine/naloxone (2/0.5, 8/2, or 16/4 mg per day). Participants will be treated for emergent withdrawal symptoms with supplemental supplemental medications (clonidine, clonazepam, compazine, ketorolac tromethamine, hydroxyzine, ranitidine, ondansetron, zolpidem) until withdrawal symptoms have dissipated, based on self-report and observer ratings. Each buprenorphine dose will be administered in equal divided doses according to a QID dosing schedule, and each dose will be maintained for a two-week period (one week of stabilization followed by one week of laboratory testing). Thus, stabilization will occur during Weeks 1, 3, and 5; testing will occur in Weeks 2, 4, and 6. Participants may receive an unaccompanied pass of up to 72 hours during Weeks 3 and 5 to attend to family obligations. Participants will be informed that urine toxicology screens will be conducted upon their return to the hospital, and that testing positive for drugs other than the study medication may result in discharge from the study. The order of administration of these three doses will vary among subjects in a randomized manner. At the completion of laboratory testing in Week 6, participants will be stabilized on 16 mg of buprenorphine. This final week of stabilization ensures that (1) any acute effects of high-dose oxycodone administration in the laboratory have dissipated and do not affect opioid dependence level; and (2) participants have sufficient opportunity to stabilize on the dose of buprenorphine on which they will be maintained during the outpatient phase.

Participants whose pain is not adequately relieved by Suboxone (buprenorphine/naloxone) will we removed from the study by the investigators. A criterion for dropout during the inpatient phase will be: clear decline in functional status, such as sustained worsening of mobility or marked decline in level of activity. In the event that average daily pain level worsens from baseline by 30% or more (e.g. 6/10 to 9/10), a clinical evaluation will be performed to consider whether the participant should be removed from the protocol, or should be allowed to continue to participate. The clinical determination will include an assessment of whether pain has improved throughout the inpatient stay as a range of doses are tested.

During the subsequent outpatient phase medication will be dispensed on a weekly basis and will consist of (1) a standing maintenance dose of 16 mg Suboxone (buprenorphine/naloxone), and (2) doses of Suboxone to be taken on a prn basis for breakthrough pain (prn doses will not exceed 25% of the total daily standing dose). Patients will report to the Substance Use Research Center (SURC) twice per week for 12 weeks for clinical visits.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV criteria for opioid abuse and prescription opioid physical dependence
2. 18-65 years of age
3. Stable weight (<10% change in 3 months) and stable physical health
4. Chronic pain syndrome (e.g., osteoarthritic pain or chronic lower back pain with/without history of surgery) of moderate (4-7) average daily pain of 6+ months duration; opioid medication maintenance for 6+ months
5. Seeking treatment for chronic pain
6. Must be expected to achieve a good analgesic effect from buprenorphine

Exclusion Criteria:

1. DSM-IV untreated Axis I disorders (e.g. MDD, BAD, psychotic disorders, eating disorders) requiring treatment
2. Regular consumption of more than 500 mg caffeine daily
3. Primary pain diagnosis of neuropathic pain, malignant pain, or headache
4. History of allergy, adverse reaction, or sensitivity to opioids, including buprenorphine
5. Pregnancy, lactation, or history of having given birth or had abortion or miscarriage within the last six months, or unwillingness to use an effective method of birth control (e.g. condoms, birth control pills, abstinence)
6. Psychotropic medications which would potentially interfere with study procedures
7. Inability to read or understand the self-report assessment forms unaided
8. Use of medications known to interfere with buprenorphine metabolism, such as disulfiram, neuroleptics, azole antifungals (e.g. ketoconazole), macrolide antibiotics (e.g. erythromycin), and HIV protease inhibitors (e.g. ritonavir, indivair, and saquinavir)
9. Methadone-dependent
10. Current heroin dependence
11. Current buprenorphine maintenance
12. History of failed treatment with buprenorphine maintenance for pain
13. Acute hepatitis with elevated liver function tests (i.e. AST and ALT > 3 times the upper limit of normal) or impaired renal function (creatinine > 1.2 )
14. Any medical condition that might interfere with the study or significantly increase the medical risks of study participation
15. Participant is currently receiving any investigational drug or has used any investigational drug within 30 days of study entry
16. History of significant cardiovascular disease, such as coronary artery disease or hypertension requiring more than two anti-hypertensive agents
17. History of insulin-dependent diabetes
18. Body mass index of <18.5 or > 35.0

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Sullivan, MD, Principal Investigator — Columbia University
Locations (1):
- SURC, New York, New York, United States

REFERENCES:
- See also: The Substance Treatment and Research Service of Columbia University (STARS) provides free and confidential treatment of substance abuse in the context of a research treatment clinical trial. — http://www.stars.columbia.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Buprenorphine/Naloxone Combination: Fifty-one (51) participants met inclusion/exclusion criteria and were randomized to a starting dose of buprenorphine/naloxone in the study (three doses were tested for 2 weeks at each dose).
Period: Randomized
Arm/Group | Buprenorphine/Naloxone Combination
Started | 51
Completed | 43 (Completed week 12)
Not Completed | 8
Period: Admission to Inpatient Phase
Arm/Group | Buprenorphine/Naloxone Combination
Started | 43
Completed | 31 (Completed 7 week inpatient phase)
Not Completed | 12
Period: 12-week Outpatient Phase
Arm/Group | Buprenorphine/Naloxone Combination
Started | 31
Completed | 18 (Completed week 12 of outpatient phase)
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Buprenorphine/Naloxone Combination
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Caucaisan | 23
  African American | 15
  Hispanic | 11
  unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Retained in Study
Description: Retention was number of participants retained at study end (Week 19).
Time Frame: week 19
Measure: Number; unit: participants
Arm/Group | Buprenorphine/Naloxone Combination
Number analyzed (Participants) | 51
participants | 18

2. Secondary Outcome: Number of Participants Abstinent From Opioids
Description: Relapse was number of participants with opioid-negative urine toxicology in last week of study participation.
Time Frame: at week 19 or length of study participation
Measure: Number; unit: participants
Groups:
- Buprenorphine/Naloxone Combination: Thirty-one (31) participants who initiated outpatient phase
Arm/Group | Buprenorphine/Naloxone Combination
Number analyzed (Participants) | 31
participants | 17

3. Secondary Outcome: Pain Measurement
Description: The primary pain measure was the Pain Assessment and Documentation Tool (PADT). Total score ranging from 0-11 reported. Higher score considered indicative of more pain. Lower score is indicative of less pain.
Time Frame: assessed twice weekly during course of 19 weeks or length of participation, only screening and last assessment reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine/Naloxone Combination
Number analyzed (Participants) | 31
units on a scale
  screening | 6.1 (1.9)
  end of study | 4.3 (0.65)

ADVERSE EVENTS:
Arm/Group | Buprenorphine/Naloxone Combination
Serious Adverse Events (participants affected / at risk) | 7/51
Other Adverse Events (participants affected / at risk) | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Buprenorphine/Naloxone Combination (N=51)
Hospitalization for rehydration/nutrition (General disorders) | 1
ER presentation for altered mental status after ingesting sleeping pills (Psychiatric disorders) | 1 — ER presentation for altered mental status after ingesting sleeping pills without self-injurious intent
cellulitis (Skin and subcutaneous tissue disorders) | 1
chest pain (Cardiac disorders) | 1
Somnolence, BP drop; intubated in ER; (General disorders) | 1
leg pain/swelling (General disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No